CLINICAL TRIAL: NCT05766683
Title: Depth of Botulinum Neurotoxin Injection for Treatment of Glabellar Lines
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David M. Ozog, Department Chair, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15627
Record Dates: First submitted 2023-02-08; First posted 2023-03-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Glabellar Frown Lines
Keywords: botulinum toxin; facial dynamic wrinkles; glabellar complex

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized using computer generated randomization list provided by PHS to either receive onabotulinumtoxinA neurotoxin injections in the glabellar complex at depth of 2mm or at depth of 4mm (or above periosteum if depth of 4mm cannot be reached)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2mm depth (Experimental): Subjects will be randomized using computer generated randomization list provided by PHS to receive onabotulinumtoxinA neurotoxin injections in the glabellar complex at depth of 2mm
  Interventions: Drug: onabotulinumtoxinA at a depth of 2mm
- 4mm depth (Experimental): Subjects will be randomized using computer generated randomization list provided by PHS to receive onabotulinumtoxinA neurotoxin injections in the glabellar complex at depth of 4mm
  Interventions: Drug: onabotulinumtoxinA at a depth of 4mm

INTERVENTIONS:
Drug: onabotulinumtoxinA at a depth of 2mm — One time administration of onabotulinumtoxinA to the corrugator supercilii muscles bilaterally. Dosing dependent on the baseline mass and volume of subject's glabellar muscles as assessed by trained cosmetic dermatologist, accounting for symmetry/asymmetry of the face and can range from 10-50 units. Will be administered at a depth of 2mm
  Arms: 2mm depth
Drug: onabotulinumtoxinA at a depth of 4mm — One time administration of onabotulinumtoxinA to the corrugator supercilii muscles bilaterally. Dosing dependent on the baseline mass and volume of subject's glabellar muscles as assessed by trained cosmetic dermatologist, accounting for symmetry/asymmetry of the face and can range from 10-50 units. Will be administered at a depth of 4mm
  Arms: 4mm depth

SUMMARY:
STUDY QUESTION: Does the depth of injection of onabotulinumtoxinA neurotoxin in the glabellar complex affect efficacy of the BoTN for the improvement of glabellar frown lines? STUDY AIM

* Primary objective: Compare the efficacy of onabotulinumtoxinA neurotoxin injected at the depth of 2mm vs 4mm for the improvement of glabellar lines
* Secondary objective: Determine any adverse effects of onabotulinumtoxinA neurotoxin injected at the depth of 2mm vs 4mm

RATIONALE FOR THE PROJECT:

Although the use of BoTN for treatment of glabellar lines has long been established as safe and effective, the optimal depth of injection has not been established. Our project hopes to establish the optimal depth of injection for onabotulinumtoxinA neurotoxin for maximal improvement of glabellar lines with minimal adverse effects

DETAILED DESCRIPTION:
STUDY AIM, BACKGROUND, AND DESIGN ABSTRACT

Botulinum neurotoxin (BoNT) is a safe and effective treatment for numerous conditions in neurology, ophthalmology, dermatology, gastroenterology, psychiatry, and urology. In dermatology, BoNT is commonly used for treatment of facial rhytides and is by far the most frequently performed cosmetic procedure in recent years. In 2002, the US Food and Drug Administration (FDA) approved the use of BoNT for the treatment of glabellar lines. Although, BoNT has shown excellent safety profile for the treatment of glabellar lines, injection methods vary widely between practitioners and no standardized method for the depth of injection has been established.

The most common treatment area is the glabellar complex, which consists of bilateral corrugator supercilii, depressor supercilii, procerus, and the orbital portion of the orbicularis oculi. With increasing age and repetitive contraction of the glabellar complex, particularly the bilateral corrugator supercilii and procerus, the formation of prominent dynamic glabellar lines and static, etched-in glabellar lines can form and lead to the appearance a more severe frown. In a study using ultrasonographic imaging and the three-dimensional scanning Cho et al. determined that the procerus was located at a depth of 3.8 ± 0.7 mm at the glabella and 2.7 ± 0.6 mm at the sellion while the intercanthal vein was located 3.0 ± 0.6 mm below the skin's surface superior to the sellion. Careful consideration of depth of injection and facial anatomy must be taken to avoid bruising and intravascular injection of BoTN. Additionally, in a cadaveric study looking at depth of corrugator supercilii of 32 Korean hemifaces using 3D scanning, Lee et al. found that the corrugator supercilii muscle rested at a depth of 5.7 +/-1.4 mm medially and 6.6 +/-1.4mm laterally and recommended BoTN injections at the depth of 4mm. However, no in vivo studies have been performed to validate this as the optimal depth of injection. In a split face study evaluating the depth of botulinum injection into the corrugator supercilii muscle no difference in brow height between injecting periosteally versus in superficial dermis. The investigators previously studied the ability of botulinum toxin to diffuse in crow's feet through laser pores into the target muscle. (8)

In our randomized study, the investigators will evaluate the efficacy of BoTN for the treatment of glabellar lines when injected at a depth of 2mm (superficial dermis) versus 4mm (intramuscularly). The investigators hypothesize that no difference exists between the two depths as the 150kD botulinum toxin molecules can easily diffuse to the target at the muscle. If this is validated, patients can be treated with more superficial depths, which will result in less pain and bruising.

STUDY HYPOTHESIS: Depth of injection of onabotulinumtoxinA neurotoxin in the glabellar complex does not affect efficacy of the BoTN for the improvement of glabellar lines.

STUDY AIM

* Primary objective: Compare the efficacy of onabotulinumtoxinA neurotoxin injected at the depth of 2mm vs 4mm for the improvement of glabellar lines
* Secondary objective: Determine any adverse effects of onabotulinumtoxinA neurotoxin injected at the depth of 2mm vs 4mm

RATIONALE FOR THE PROJECT:

Although the use of BoTN for treatment of glabellar lines has long been established as safe and effective, the optimal depth of injection has not been established. Our project hopes to establish the optimal depth of injection for onabotulinumtoxinA neurotoxin for maximal improvement of glabellar lines with minimal adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18 and older
2. Patient able to understand requirements of the study and risks involved
3. Patient able to sign a consent form

Exclusion Criteria:

1. A patient who is lactating, pregnant, or planning to become pregnant
2. Prior history of botulinum neurotoxin treatment of the face within the past one (1) year
3. History of hypersensitivity to botulinum neurotoxin
4. History of neuromuscular disorders (e.g., myasthenia gravis)
5. History of facial surgery or scars in the treatment area that may confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Injection of onabotulinumtoxinA, 2 mm depth | 120 days
  Assess the efficacy of onabotulinumtoxinA neurotoxin injected at the depth of 2mm for the improvement of glabellar lines using the Merz aesthetics scales.
  The Merz scale is as follows:
  0 - no glabellar lines
  1- mild glabellar lines 2 - moderate glabellar lines 3 - severe glabellar lines 4 - very severe glabellar lines
Injection of onabotulinumtoxinA, 4 mm depth | 120 days
  Assess the efficacy of onabotulinumtoxinA neurotoxin injected at the depth of 4mm for the improvement of glabellar lines using the Merz aesthetics scales.
  The Merz scale is as follows:
  0 - no glabellar lines
  1- mild glabellar lines 2 - moderate glabellar lines 3 - severe glabellar lines 4 - very severe glabellar lines

SECONDARY OUTCOMES:
Secondary Outcome Measure | 120 days
  Incidence of any adverse effects of onabotulinumtoxinA neurotoxin injected at the depth of 2mm vs 4mm.
Efficacy comparison | 120 days
  Compare the efficacy of onabotulinumtoxinA neurotoxin injected at the depth of 2mm vs 4mm for the improvement of glabellar lines using the Merz aesthetics scale.
  The Merz scale is as follows:
  0 - no glabellar lines
  1- mild glabellar lines 2 - moderate glabellar lines 3 - severe glabellar lines 4 - very severe glabellar lines

CONTACTS AND LOCATIONS:
Overall Officials: David Ozog, MD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Giordano CN, Matarasso SL, Ozog DM. Injectable and topical neurotoxins in dermatology: Indications, adverse events, and controversies. J Am Acad Dermatol. 2017 Jun;76(6):1027-1042. doi: 10.1016/j.jaad.2016.11.012. PMID 28522039
- [Background] Gostimir M, Liou V, Yoon MK. Safety of Botulinum Toxin A Injections for Facial Rejuvenation: A Meta-Analysis of 9,669 Patients. Ophthalmic Plast Reconstr Surg. 2023 Jan-Feb 01;39(1):13-25. doi: 10.1097/IOP.0000000000002169. Epub 2022 Mar 30. PMID 35353777
- [Background] Giordano CN, Matarasso SL, Ozog DM. Injectable and topical neurotoxins in dermatology: Basic science, anatomy, and therapeutic agents. J Am Acad Dermatol. 2017 Jun;76(6):1013-1024. doi: 10.1016/j.jaad.2016.11.022. PMID 28522038
- [Background] Cho Y, Lee HJ, Lee KW, Lee KL, Kang JS, Kim HJ. Ultrasonographic and Three-Dimensional Analyses at the Glabella and Radix of the Nose for Botulinum Neurotoxin Injection Procedures into the Procerus Muscle. Toxins (Basel). 2019 Sep 24;11(10):560. doi: 10.3390/toxins11100560. PMID 31554222
- [Background] Lee HJ, Lee KW, Tansatit T, Kim HJ. Three-Dimensional Territory and Depth of the Corrugator Supercilii: Application to Botulinum Neurotoxin Injection. Clin Anat. 2020 Jul;33(5):795-803. doi: 10.1002/ca.23507. Epub 2019 Nov 13. PMID 31637771
- [Background] Sneath J, Humphrey S, Carruthers A, Carruthers J. Injecting botulinum toxin at different depths is not effective for the correction of eyebrow asymmetry. Dermatol Surg. 2015 Jan;41 Suppl 1:S82-7. doi: 10.1097/DSS.0000000000000159. PMID 25548850
- [Background] Mahmoud BH, Burnett C, Ozog D. Prospective randomized controlled study to determine the effect of topical application of botulinum toxin A for crow's feet after treatment with ablative fractional CO2 laser. Dermatol Surg. 2015 Jan;41 Suppl 1:S75-81. doi: 10.1097/01.DSS.0000452642.83894.ab. PMID 25548849